CLINICAL TRIAL: NCT02777697
Title: Cancer Chronic Pain Predicted by Emotional and Cognitive Status
Acronym: CanoPEe
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0262
Record Dates: First submitted 2016-04-13; First posted 2016-05-19 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2016-05

CONDITIONS: Chronic Pain; Cancer
Keywords: cancer treatment protocols; chronic cancer pain; cognitive function; quality of life; anxiety; depression
MeSH Terms: conditions — Chronic Pain; Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- cancer patients
  Interventions: Other: chronic pain

INTERVENTIONS:
Other: chronic pain

SUMMARY:
The aim of this study is to investigate the predictive dimension of cognitive-emotional status of cancer patients on the chronic pain development 6 months after different cancer treatment protocol (surgery, chemotherapy, radiotherapy, hormone therapy, targeted therapy ...).

DETAILED DESCRIPTION:
This is an observational, longitudinal and multicenter study assessing in cancer patients the link between the cognitive-emotional status and the development of chronic pain.

Cognition, anxiety, depression, quality of life, social vulnerability, cancer perception, pain and analgesic consumption are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Cancer patient with one or more programmed cancer treatment protocols (chemotherapy, surgery, hormone therapy, radiation therapy, targeted therapy, ...)
* Acceptance to sign the non-opposition form

Exclusion Criteria:

* History of cancer and cancer treatment protocols (chemotherapy, surgery, hormone therapy, radiation therapy, targeted therapy, ...)
* History and/or presence of primary brain tumors (glioblastoma, meningioma, neurofibroma ...)
* History of neurological disorders (Parkinson's disease, Alzheimer's disease, dementia, epilepsy, moderate to severe head injury, ...)
* History of psychiatric disorders (schizophrenia, bipolar disorder, ...)
* Medical and surgical history incompatible with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Measure of average pain intensity by a numerical rating scale | 7 days before the visit
  Measure of average pain intensity by a numerical rating scale assessed 7 days before the 6 months visit after inclusion of patients.

SECONDARY OUTCOMES:
Pain assessment by numerical rating scale and DN4 | at baseline
Pain assessment by numerical rating scale and DN4 | at 6 months
Pain assessment by numerical rating scale and DN4 | at 12 months
Pain assessment by numerical rating scale and DN4 | at 24 months
Pain assessment by numerical rating scale and DN4 | 2 days after each cancer treatment protocol
Evaluation of analgesic consumption | at day 1
  Analgesic consumption is evaluated during all period of the study (name of the specialty, dose, indication, form, administration route, starting date, end date),
Cognitive assessment by Trail Making Test A and B (TMT) | at baseline
Cognitive assessment by Trail Making Test A and B (TMT) | at 24 months
Cognitive assessment by Trail Making Test A and B (TMT) | at 6 months
Cognitive assessment by Trail Making Test A and B (TMT) | at 12 months
Rey Auditory-Verbal Learning Test (RAVLT) and FACT-COG | at baseline
Rey Auditory-Verbal Learning Test (RAVLT) and FACT-COG | at 24 months
Rey Auditory-Verbal Learning Test (RAVLT) and FACT-COG | at 12 months
Rey Auditory-Verbal Learning Test (RAVLT) and FACT-COG | at 6 months
Quality of life assessment | at baseline, 6 months, 12 months and 24 months,
  Quality of life assessment by:
  - The European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30), at baseline, 6 months, 12 months and 24 months. This questionnaire assesses the quality of life of cancer patients. It is divided in 9 subscales consisting of several items: 5 subscales measuring functional status (physical, role, social, emotional, cognitive), three subscales measuring symptoms (fatigue, pain, nausea and vomiting) and a global subscale of quality of life and health. Finally, six items/isolated symptoms, covering cancer symptoms and frequent side effects of cancer therapies (e.g. loss of appetite) are also included in the EORTC QLQ-C30. The EORTC QLQ-C30 Score ranges from 0 to 126
Social vulnerability assessment by EPICES questionnaire | at baseline, 6 months, 12 months and 24 months
Anxiety and Depression assessment by HAD scale | at baseline, 6 months, 12 months and 24 months
Illness perception assessment | at baseline, 6 months, 12 months and 24 months
  Global score ranges from 0 to 200
Coping strategies assessment by Coping strategies questionnaire (CSQ) | 2 days after each cancer treatment protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France